CLINICAL TRIAL: NCT06419881
Title: Tele-Drama Therapy for Community-Dwelling Older Adults With Constricted Life Space Mobility: A Mixed Methods Randomized Control Study
Brief Title: Tele-Drama Therapy for Community-Dwelling Older Adults With Constricted Life Space Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Uniper Care (Unknown)
Responsible Party: Principal Investigator, Shoshi Keisari, Principal Investigator, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 217/22
Record Dates: First submitted 2024-05-09; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Constricted Life Space Mobility; Tele-drama Therapy
Keywords: Life Space Mobility; Tele-drama therapy intervention; Older Adults; Mental health; Social Connectedness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to eight tele-drama therapy treatment groups or eight usual care groups. Participants in the experiment group received a 12-week tele-drama therapy intervention, with each session lasting 75 minutes via the Uniper Care platform. Participants in the usual care groups continued to receive the routine activities provided by Uniper Care. As a token of gratitude for their participation, participants in the control groups were offered a 3-session online playback theater workshop, in addition to a gift card.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-drama therapy intervention (Experimental): This arm received a 12-week tele-drama therapy intervention, with each session lasting 75 minutes via the Uniper Care platform.
  Interventions: Behavioral: Tele-drama therapy
- Usual Care (Other): This usual care arm continued to receive routine activities provided by Uniper Care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Tele-drama therapy — A 12-week tele-drama therapy group intervention integrating Playback Theater and Life Review Therapy
  Arms: Tele-drama therapy intervention
Other: Usual Care — This arm continued to receive the routine activities provided by Uniper Care
  Arms: Usual Care

SUMMARY:
Older adults with constricted life-space mobility face increased risk of social isolation and poor mental health. Despite the benefits of therapeutic interventions, the literature indicates low use of mental health services in the older population, often due to mobility limitations and/or negative attitudes toward psychotherapy. Developing accessible interventions that address negative attitudes towards mental health services is crucial. Group drama therapy has shown to improve the mental health of older adults, and the creative process itself may help overcome stigmas associated with seeking mental health services. The aim of this study was to explore a 12-week tele-drama therapy group intervention tailored for older adults with constricted mobility. The intervention integrated playback theatre and life review therapy, and was delivered via Uniper Care, an accessible technology designed for older adults. The study will explore the contribution of the intervention and will examine the relationship between processes in drama therapy and their contribution on older adults mental health. This study will also explore the experience of participants, therapists and staff members.

DETAILED DESCRIPTION:
Older adults suffering from constricted life space mobility experience higher rates of chronic disease, functional and cognitive impairments, depressive symptoms, limited access to medical care and minimal social encounters. Interventions that enhance social skills and increase opportunities for social interaction have showed promising results, but for older adults with constricted life space mobility, this is especially challenging since access to social encounters is limited. Tele-therapy offers a potential solution to these physical barriers and have been proven effective in treating common mental disorders, such as anxiety. However, a recent tele-therapy study that found that while participants appreciated the possibility of online therapy, many still refused to participate because they were not interested in focusing on sensitive subjects, such as their depression. These findings highlight the crucial need to develop accessible interventions that address these potential physical and emotional barriers that may prevent older adults with constricted mobility from consuming mental health services. Tele-drama therapy can offer a solution to these barriers, however the unexplored potential of online group drama therapy with older adults remains.

The aim of this Randomized Control, mixed methods study was to explore a 12-week tele-drama therapy group intervention tailored for older adults with constricted mobility. The quantitative arm of this mixed-methods study aims to examine the impact of a tele-drama therapy intervention on the mental health of older adults with constricted life space mobility, and to pinpoint the associations between dramatic processes and outcome measures. The researchers hypothesize that Tele-drama therapy will (1) enhance social connectedness, self-acceptance, personal growth, and a sense of meaning in life, as compared to the control condition, (2) reduce depressive symptom and loneliness as compared to the control condition. In addition, the researchers hypothesize that in-session therapeutic change factors will predict better outcomes in the treatment group.

The qualitative arm of this study will explore the experiences of participants and staff members.

Participants:

This study aimed to recruit 120 participants, factoring in a 15% dropout rate, based on an a-priori power analysis. The intervention was offered to 3,595 Uniper Care members residing throughout Israel. Participants were recruited over eight months and were randomly assigned to eight tele-drama therapy treatment groups or eight usual care groups who continued to receive the routine activities provided by Uniper Care.

A total of 111 participants completed the study (88 % of those who started the intervention): 51 from the experimental groups and 60 from the control groups. A total of 15 participants (11.9%) dropped out throughout the study.

The Online Platform:

Uniper Care is a social club aimed to promote active aging using accessible technology designed with and for older adults. Uniper Care's service is delivered via the TV by connecting a remote and a camera to any TV that turns the TV from passive to interactive. Uniper Care is also accessible via other digital devices such as tablets, smart phone and desktop. Uniper Cares' service includes daily classes around physical, social, emotional and cognitive well-being, along with recorded programs and videos and gamification of various training.

The Tele-drama Therapy Group Intervention:

Eight groups of up to eight participants received a 12-week tele-drama therapy intervention, with each session lasting 75 minutes via the Uniper Care platform Sessions were delivered by four certified drama therapists who received training on the treatment protocol before the intervention. All sessions were recorded using OBS (Open Broadcast Software, v29.0.0) an external software program for screen recording and live streaming. All the recordings were secured on a computer with a password for further coding of the data.

The 12-week intervention consisted of four stages: (1) Introduction (sessions 1-2): establishing participant acquaintance, a therapeutic alliance and a safe space for self-expression and exploration, (2) Life-review on stage (sessions 3-8): revisiting past positive life stories from new viewpoints, (3) Looking ahead (sessions 9-11): exploring future stories and goals to foster a sense of purpose and sense of self-development, and (4) Farewell: reflecting upon the group process and achievements, and closure.

Measures:

A demographic questionnaire administered at baseline.

Outcome measures were assessed pre and post intervention for all participants. Process measures were assessed for participants in the experimental groups after session No. 10.

Control variables (individual traits/differences) were assessed at baseline to examine their potential role as covariates.

Semi-structured interviews were held with participants from three experimental groups, three drama therapists, and two Uniper Care community coordinators. The interviews were recorded and transcribed for further coding and analysis.

Data Analysis:

Quantitative Analysis:

Statistical data will be collected and analyzed in SPSS, version 27, and R, version 3.5.

The reliability of the study's scales will be assessed using Cronbach's alpha for internal consistency.

Shapiro-Wilk test of normality will be conducted to determine whether the outcome variables are normally distributed.

Chi square, t-tests or one-way ANOVA to examine differences between variables and groups, and some additional variables.

Correlations will be calculated to analyze the relationships between sociodemographic, control, and outcome variables.

To examine the effects of the intervention on outcome variables, the analysis will include repeated measures (pre/post) with mixed-models (random effects) by groups (Experiment/Control) including interaction between time X groups.

Further follow-up exploratory analyses will attempt to find associations between outcome and process variables and individual traits.

Qualitative Analysis:

To explore the experiences of participants and staff members, qualitative analysis of the semi-structured interviews will apply reflexive thematic analysis of interviews (Braun & Clarke, 2019).

ELIGIBILITY:
Inclusion Criteria:

1. age 65 and over with constricted life space mobility
2. with normal cognitive functioning (assessed by the research coordinator and community coordinators at Uniper Care)
3. selected by the research coordinator and community coordinators as suitable to participate in a treatment group
4. with sufficient mastery of the Hebrew language
5. with an absence of a diagnosis of a mental disorder
6. who expressed interest in taking part in a drama therapy intervention and provided informed consent.

Exclusion Criteria:

1. older adults who experienced the loss of a souse or child six months prior to the intervention
2. participants in the experimental group who missed four or more of the 12 sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-01-29 (Actual)

PRIMARY OUTCOMES:
Social Connectedness | (1) Baseline, (2) Post intervention
  Social connectedness was measured using a composite score of two measures: The 10-item satisfaction in social relationships subscale from the UCLA loneliness scale (Russell et al., 1980), and the 9-item positive relationships with others subscale of the psychological well-being scale (Ryff, 1991); both measures were rated on a 5-point scale.
Psychological well-being | (1) Baseline, (2) up to 1 week post intervention
  Psychological well-being was measured using two subscales from the Ryff scale (1991): self-acceptance and personal developement , which were rated from 1 (Strongly disagree) to 5 (Strongly agree).
Meaning in life | (1) Baseline, (2) up to 1 week post intervention
  Meaning in life was measured using an abridged 8-items version (Krause, 2007), adapted for older adults. Items were rated from 1 (Strongly disagree) to 5 (Strongly agree).
Well-being | (1) Baseline, (2) up to 1 week post intervention
  Well-being was measured using the 5-item WHO-5 scale (Gosling et al., 2003; Keisari et al., 2022). Items were rated from 0 (Never) to 5 (All the time).
Loneliness | (1) Baseline, (2) up to 1 week post intervention
  Loneliness was measured using the 10-item dissatisfaction in social relationships subscale from the UCLA loneliness scale (Russell et al., 1980), with an additional item ("I feel lonely"). Items were rated from 1 (Never) to 5 (Always).
Depressive symptoms | (1) Baseline, (2) up to 1 week post intervention
  Depressive symptoms were measured using the Geriatric Depression Scale (Yesavage et al., 1982), a questionnaire composed of 15 yes/no questions that relate to how participants felt in the previous week.

SECONDARY OUTCOMES:
Therapeutic alliance | up to 1 week after session No. 10
  Therapeutic alliance was measured using a 17-item alliance in art therapy questionnaire (Bat Or & Zilcha-Mano, 2018), which was slightly adapted to the field of drama therapy by the research team. Items were rated from 1 (Does not describe my experience at all) to 5 (Completely describes my experience.
Meaningfulness in drama therapy | up to 1 week after session No. 10
  Meaningfulness in drama therapy was measured using a 15-item questionnaire (Baker et al., 2016), which was slightly adapted to measure the extent of meaning experienced by participants in the drama therapy process. Items were rated from 1 (Does not describe my experience at all) to 5 (Completely describes my experience.
Vitality | up to 1 week after session No. 10
  Vitality was measured using a 5-item questionnaire that measured the subjective experience of feeling vital during the drama therapy session prior to the questionnaire (Ryan & Frederick, 1997). Items were rated from 1 (Does not describe my experience at all) to 5 (Completely describes my experience.
Subjective social support | up to 1 week after session No. 10
  Subjective social support was measured using the 6 items from the abbreviated Duke social support index questionnaire (Koenig et al., 1993), with "family and friends" changed to "group members.". Items were rated from 1 (Hardly ever) to 3 (Most of the time
Flow | up to 1 week after session No. 10
  Flow was measured using the 7-item state flow scale (Martin & Jackson, 2008). Items were rated from (Does not describe my experience at all) to 5 (Completely describes my experience).
Client involvement in group drama therapy - Therapists assessment | up to 1 week post intervention
  This measure of Client involvement in group drama therapy was assessed by drama therapists who rated a single-item question: "for each participant in the group, think about the way he/she behaved in the group and rate the extent of his/her active involvement in the dramatic process of treatment", from 1 ((Not at all) to 5 (Completely)).
Client involvement in group drama therapy - Investigators assessment | up to 1 week post intervention
  This measure of Client involvement in group drama therapy was assessed by one of the research investigators using the 11-item Client Involvement and Interaction in Group DT (Tobon et al., 2011), an observational rating scale that was completed for each participant based on video recordings of three tele-DT sessions (2, 6, and 11). Items (were rated from 0 (never present) to 4 (always present

CONTACTS AND LOCATIONS:
Overall Officials: Shoshi Keisari, PhD, Principal Investigator — University of Haifa; Hod Orkibi, PhD, Principal Investigator — University of Haifa
Locations (1):
- Uniper Care, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Yes
Upon Request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after publication
Access Criteria: Upon Request